CLINICAL TRIAL: NCT01376050
Title: A Double-Blind, Placebo-Controlled Randomized Evaluation of the Effect of the Erchonia ML Scanner (MLS) on Venous Stasis Ulcers
Brief Title: Efficacy Study of the Application of Low Level Laser Light to Treat Venous Stasis Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC_VSU
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Venous Stasis Ulcer
Keywords: venous stasis ulcer; leg ulcer
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erchonia ML Scanner (MLS) (Active Comparator): Erchonia MLS comprises three 17.5 milliWatts (mW) 635 nanometer (nm) light emitting diodes. The center diode is fixed at 6 inches above the venous stasis ulcer center, and the other 2 diodes rotate about this center fixed diode for 20 minutes. Total dosage delivered to the skin is 2.95 J/cm squared.
  Interventions: Device: Erchonia ML Scanner (MLS)
- Placebo Laser (Placebo Comparator): Placebo Laser has the same appearance and application as the Erchonia MLS but does not emit an therapeutic output.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia ML Scanner (MLS) — Erchonia MLS comprises three 17.5 mW 635 nm diodes. The center diode is fixed at 6 inches above the venous stasis ulcer center and the other 2 diodes rotate about this center fixed diode for 20 minutes. Total dosage delivered to the skin is 2.95 J/cm squared.
  Arms: Erchonia ML Scanner (MLS)
Device: Placebo Laser — Placebo Laser has no therapeutic output emitted.
  Arms: Placebo Laser

SUMMARY:
The purpose of this study is to determine whether low level laser light therapy is effective as an adjunctive therapy to the healing of venous stasis leg ulcers.

DETAILED DESCRIPTION:
A chronic venous stasis leg ulcer is a wound below the knee that fails to heal within 6 weeks. Venous stasis ulcers account for 80% to 90% of all leg and foot ulcers, affecting an estimated 500,000-600,000 people in the United States every year. Venous stasis ulcers account for the loss of 2 million working days and incur treatment costs around $3 billion dollars annually in the United States. Standard of care for venous stasis ulcers includes compression of the affected leg together with daily dressing changes to minimize swelling; debridement of the ulcer to remove dead tissue and bacteria; and daily wound Care dressing to keep the wound clean. Venous stasis ulcers typically have very lengthy and poor healing rates, with up to 50% remaining open and unhealed for 9 months or longer. Many patients suffer pain and sleep and mobility problems, impairing quality of life. Recurrence rates for venous stasis ulcers is very high, with about one third of treated individuals experiencing 4 or more episodes of ulceration.

Low level laser light therapy (LLLT), with its proven tissue healing acceleration properties has recently gained attention as a simple, non-invasive alternative adjunctive therapy to assist in both wound closure and accelerated time to wound closure. Numerous histological trials have exhibited laser therapy's capacity to upregulate essential wound-healing factors such as vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), oxygen concentration, fibroblast proliferation, collagen synthesis, re-epithelialization, and tissue granulation. Clinically, the application of laser therapy has demonstrated promise, accelerating the rate of wound healing and tissue contracture.

ELIGIBILITY:
Inclusion Criteria:

* At least one venous stasis ulcer, diagnosed according to a differential diagnosis methodology that satisfies both criteria supportive of the ulcer's venous origin and criteria that eliminates the ulcer as being indicative of non-venous origin. Diagnostic criteria to evaluate satisfaction of criteria that is supportive of venous origin of the ulcer will involve an evaluation of medical history and wound history variables; physical examination of the affected leg and ulcer site; and objective testing
* Resting Ankle Brachial Pressure Index (ABPI) of 0.8 or greater
* Venous Doppler ultrasound shows reflux in the suspect vein
* Clinical Etiologic Anatomic Pathophysiologic (CEAP) Classification System Class 6
* Ulcer measures 5 to 20cm², inclusive, according to standardized computerized planimetry evaluation
* presenting venous leg ulcer has been present for 6 continuous weeks or longer
* Subject agrees to not partake in any other form of treatment for the ulcer throughout study participation, other than the standard of care treatment provided by the investigator as part of the study protocol

Exclusion Criteria:

* Satisfaction of any exclusive diagnostic criteria that is considered indicative of an ulcer being of non-venous origin (e.g. arterial or mixed origin), or as having a non-venous component. This evaluation will include consideration of medical history and wound history variables; examination of the affected leg and ulcer site; and objective tests and measurements
* Resting Ankle Brachial Pressure Index (ABPI) of less than 0.8
* Doppler ultrasound that shows absence of reflux in the suspect vein
* Fasting blood glucose (blood sugar) level of greater than 140 mg/dl that is indicative of current or potential diabetes
* Subject presents with factors that may significantly impede or delay the healing of chronic non-healing wounds, including known diabetes or other disordered glucose metabolic disease; malnutrition; collagen diseases such as Ehlers-Danlos syndrome; history of systematic glucocorticosteroid therapy; history of exogenous glucocorticosteroid therapy; and chemotherapeutic (antineoplastic) drug use
* Ulcer has significant bacterial infection, confirmed by a positive swab culture utilizing Levine's technique
* Ulcer has been present for less than 6 continuous weeks
* Ulcer is of CEAP Class 0 through 5, inclusive
* Ulcer measures less than 5cm² or greater than 20cm², according to standardized computerized planimetry evaluation
* Exposed bone tendon or fascia
* General skin disorder such as psoriasis or penicilitis
* Immunosuppressive disorder
* Hypercoagulable state
* Prior deep vein thrombosis
* Cellulites during the one-year period prior to study participation in
* Vasculitis or collagen vascular disease
* History of prior venous surgery
* Any concomitant illness(es) or medical condition(s) that would render the subject inappropriate for the study (i.e., renal failure, liver disease, connective tissue disorders, etc.)
* Active or recurrent cancer or currently receiving chemotherapy or radiation therapy
* Subject is taking a regimen of any medication(s) that may affect wound healing, including corticosteroid, chemotherapeutic and non-steroidal anti-inflammatory (NSAID) medications
* Developmental disability/significant psychological disorder that could impair the subject's ability to provide informed consent, participate in the study protocol or record study measures, including schizophrenia, bipolar disorder and psychiatric hospitalization within the last 2 years
* Females currently pregnant or lactating or intending to attempt to become pregnant during the course of intended study participation
* Involvement in litigation/receiving disability benefits related to venous stasis ulcer(s).
* Other research participation in the 30 days prior to study qualification evaluation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Kenkel, MD, Principal Investigator
Locations (2):
- Jeffrey Kenkel, MD, Dallas, Texas, United States
- Luc Teot, MD, Montpellier, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Erchonia ML Scanner (MLS): Erchonia ML Scanner (MLS) comprises three 17.5 milliWatts (mW) 635 nanometer (nm) light-emitting diodes. The center diode is fixed at 6 inches above the venous stasis ulcer center and the other 2 diodes rotate about this center fixed diode for 20 minutes. Total dosage delivered to the skin is 2.95 J/cm squared.
- Placebo Laser: Placebo Laser has the same appearance and function as the Erchonia MLS but not does emit any therapeutic output.
Period: Overall Study
Arm/Group | Erchonia ML Scanner (MLS) | Placebo Laser
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erchonia ML Scanner (MLS) | Placebo Laser | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.92 (14.78) | 65.80 (11.17) | 67.00 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 13 | 11 | 24
Ulcer Size [Mean (Standard Deviation); unit: cm²] — The study ulcer was digitally photographed, and the ulcer size/area calculated in centimeters squared (cm²) using the Aranz Medical SilhouetteMobile™ System, a portable handheld computer device with custom camera and software that enables capturing of a wound image at the point of care.
  cm² | 10.13 (6.23) | 11.30 (7.55) | 10.53 (6.64)
Visual Analog Scale (VAS) Degree of Ulcer Pain Rating [Mean (Standard Deviation); unit: units on a scale] — The Visual Analog Pain Scale (VAS) is one of the three most commonly used scales for assessing pain. The VAS scale ranges from 0 to 100 mm, with 0 indicating no pain and 100 indicating worst pain imaginable. The subject marks on the line the spot for the pain intensity, which is then measured. Subjects in this study were asked to mark the spot on the line that best represented the degree of pain they felt at the study ulcer site at that time.
  units on a scale | 44.69 (23.93) | 30.45 (20.04) | 38.17 (22.93)

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Proportion of Venous Stasis Ulcers Attaining Complete Wound Closure Between Treatment Groups
Description: 'Complete wound closure' is defined as skin re-epithelialization without drainage or dressing requirements confirmed across a consecutive two-week evaluation period. Efficacy success was defined as a statistically significant greater proportion of venous stasis ulcers in the test procedure group achieving complete wound closure compared with the proportion of venous stasis ulcers in the placebo procedure group achieving complete wound closure.
Time Frame: Baseline and 12 Weeks
Measure: Number; unit: participants
Arm/Group | Erchonia ML Scanner (MLS) | Placebo Laser
Number analyzed (Participants) | 13 | 11
participants | 3 | 2
Statistical Analysis 1: Comparison: Erchonia ML Scanner (MLS) vs Placebo Laser; Test type: Superiority or Other; p > 0.05, Fisher Exact

2. Secondary Outcome: Change in Ulcer Size
Description: The study ulcer was digitally photographed, and the ulcer size/area calculated in centimeters squared (cm²) using the Aranz Medical SilhouetteMobile™ System, a portable handheld computer device with custom camera and software that enables capturing of a wound image at the point of care. The change in ulcer size from baseline to study endpoint (12 weeks) was calculated. A decrease in ulcer size indicates an improvement in the ulcer status and is positive for study success. An increase in ulcer size indicates a worsening of the ulcer status and is negative for study success.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | Erchonia ML Scanner (MLS) | Placebo Laser
Number analyzed (Participants) | 13 | 11
cm² | -6.26 (3.66) | -6.72 (5.06)
Statistical Analysis 1: Comparison: Erchonia ML Scanner (MLS) vs Placebo Laser; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 13 Weeks
Arm/Group | Erchonia ML Scanner (MLS) | Placebo Laser
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No